CLINICAL TRIAL: NCT02977663
Title: Imaging Multiparametric/Multimodality (Magnetic Resonance Imaging Combined With Positron Emission Tomography) for Lungcancer
Brief Title: Imaging Multiparametric/Multimodality for Lungcancer
Acronym: IRMomics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: General Electric (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: K160701; ANSM (Registry Identifier: N° ID RCB : 2016-A00813-48)
Record Dates: First submitted 2016-11-10; First posted 2016-11-30 (Estimated); Last update posted 2021-01-08 (Actual); Status verified 2020-12

CONDITIONS: Lungcancer
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnetic Resonance Imaging (MRI) (Other): Thoracic Magnetic Resonance Imaging (MRI)
  Interventions: Other: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Other: Magnetic Resonance Imaging (MRI) — * Chest MRI during the MRI cerebral
  * 2 tubes of blood taken during the medical visit

SUMMARY:
1. To build an imaging biobank of 200 patients with lungcancer, including pathologic and molecular characteristics of the tumor (mutational status, circulating DeoxyriboNucleic Acid (DNA) from serum biobank…), staging of the cancer (according to the new 2016 Tumor Node Metastasis (TNM) status, the table that classify non-small cell lungcancer) and follow-up informations (Response to first-line treatment (Response Evaluation Criteria in Solid Tumors (RECIST)), disease-free survival, 1-3 years survival).
2. To propose a simple severity scoring system based on tumor features such as size, doubling time (if available), location, amount of enhancement and necrosis. Such approach has been proposed for glioma evaluation (Visually Accessible Rembrandt Images (VASARI)) but is not available for the lung. The objective is to do better than the Tumor Node Metastasis (TNM) staging.
3. To develop and evaluate an IntraVoxel Incoherent Motion (IVIM) protocol for lungcancer evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years
* High suspicion of lungcancer confirmed
* Tumor > 2 cm
* Incomplete cerebral staging or not yet realized in the initial consultation of screening

Exclusion Criteria:

* Lungcancer medical history
* During Pregnancy
* Contraindications to MRI
* Patient not able to understand the information of the protocol, taking into account the state of the brain
* Patient unable to keep lying in MRI the necessary time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-08-28 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Event-free survival of patients with lungcancer | 3 years

SECONDARY OUTCOMES:
Overall survival | 3 months, 1 year, 2 years and 3 years
Number of patients by histologic subtypes | 3 months, 1 year, 2 years and 3 years
Number of patients by mutational profile | 3 months, 1 year, 2 years and 3 years
Number of patients with metastases | 3 months, 1 year, 2 years and 3 years
Number of patients with brain metastases | 3 months, 1 year, 2 years and 3 years
Number of metastases by patient | 3 months, 1 year, 2 years and 3 years
Therapeutic responses assessed by scanner/MRI and/or Positron Emission Tomography (PET) based on consensus criteria (RECIST 1.1 and PET Response Criteria in Solid Tumors (PERCIST)) | 3 months, 1 year, 2 years and 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- BRILLET, Bobigny, France

IPD SHARING:
Plan to Share IPD: No